CLINICAL TRIAL: NCT05839925
Title: Prevalence of Temporomandibular Joint Dysfunction in Patients With Ankylosing Spondylitis and Comparison of the Findings With Healthy Controls
Brief Title: Prevalence of Temporomandibular Joint Dysfunction in Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstanbulPRMTRH
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Temporomandibular Joint Disorders; Temporomandibular Disorders; TMJ; Spondyloarthropathy
MeSH Terms: conditions — Spondylitis, Ankylosing; Temporomandibular Joint Disorders; Spondylarthropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankylosing spondylitis group: The patients were selected on a randomized form among the patients with a diagnosis of AS according to the modified New York criteria who referred to Istanbul Physical Medicine Rehabilitation Training and Research Hospital.
  Interventions: Diagnostic Test: Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) Axis I and II
- Healthy volunteers: Healthy volunteers between the ages of 18-75 were selected randomly.
  Interventions: Diagnostic Test: Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) Axis I and II

INTERVENTIONS:
Diagnostic Test: Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) Axis I and II — The presence of temporomandibular joint dysfunction was evaluated using the diagnostic criteria for temporomandibular disorders (DC/TMD).

SUMMARY:
This study included 113 patients diagnosed with ankylosing spondylitis and 110 healthy volunteers. Participants in both groups were evaluated using the 'Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)' diagnostic criteria. In addition, the relationship between temporomandibular joint dysfunction and disease activity was investigated in patients with ankylosing spondylitis.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic, inflammatory disease with an unknown etiology that primarily affects the axial spine, especially the sacroiliac joints, and can also involve peripheral joints and extra-articular clinical manifestations. Complaints related to temporomandibular joint pathologies are commonly observed in the general population but more frequent in the group of patients diagnosed with ankylosing spondylitis compared to the average population. Although the mechanism of temporomandibular joint involvement in ankylosing spondylitis is not fully understood, destruction of the joint capsule or disk, synovitis in the joint, and craniovertebral postural changes have been suggested as possible mechanisms. In addition, pain due to temporomandibular joint dysfunction can significantly affect daily life activities, quality of life, social participation, and the emotional status of the individual. Determining the level of relationship between quality of life and psychological status will support the development of new interventions and treatment approaches to improve patient's quality of life further.

The age, gender, body mass index, marital status, duration of ankylosing spondylitis (AS) diagnosis, symptom onset, treatment for AS, occupation, smoking status, and Human Leukocyte Antigen (HLA)-B27 positivity status were recorded for the patient. The 'Diagnostic Criteria for Temporomandibular Disorders (DC/TMD),' published in 2014 and translated into Turkish in 2016, was used to assess the presence of temporomandibular joint dysfunction in the patients. This evaluation system consists of two parts: the clinical evaluation and examination findings of the current pathology on Axis I, and the psychosocial status of the disease on Axis II. The questions in the Symptom Questionnaire on the first axis were directed to the patient, and then the results were recorded by performing the examinations indicated on the examination form. The diagnosis was determined according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) decision tree, and marked on the examination form. Two groups were created based on the decision tree: pain and joint disorders. Pain disorders were further subdivided into muscle pain, joint pain, and TMD-related headaches; muscle pain was further subdivided into local muscle pain, muscle-fascial pain, and referred muscle-fascial pain subgroups. Joint disorders were classified as disc displacement with reduction, disc displacement with reduction-intermittent locking, disc displacement without reduction-limited mouth opening, disc displacement without reduction-limited mouth opening, degenerative joint disease, and dislocation.

On Axis II, the patients were asked to mark the areas where they felt pain on the pain drawing form. The marked area was divided into categories according to its size. The level of experienced pain was evaluated with the Graded Chronic Pain Scale (GCPS), jaw function limitations were assessed with the Jaw Functional Limitation Scale-20 (JFLS-20), depression was evaluated with the Patient Health Questionnaire-9 (PHQ-9), anxiety was assessed with the General Anxiety Disorder 7 (GAD-7), physical symptoms were evaluated with the Patient Health Questionnaire-15 (PHQ-15), and parafunctional activities were evaluated with the Oral Behavior Checklist (OBC). Additionally, the relationship between the identified diagnosis and psychosocial factors, disease activity, and other disease-specific factors was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Ankylosing Spondylitis according to the Modified New York Criteria between the ages of 18-75.
* Healthy volunteers between the ages of 18 and 75.

Exclusion Criteria:

* Changes in the treatment of ankylosing spondylitis within the last 6 months
* Patients with pathology related to the temporomandibular joint and associated structures prior to the diagnosis of ankylosing spondylitis
* Use of medication that affects bone metabolism
* Presence of neurological or cognitive deficits
* History of trauma, malignancy, infection, and surgery in the head and neck area
* Presence of dental or periodontal pain
* History of orthodontic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 113 patients with ankylosing spondylitis were diagnosed and 110 healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) Axis I Symptom questionnaire | A single point in time (1 day)
  The presence of temporomandibular joint dysfunction will be evaluated using the The questionnaire that investigates temporomandibular region pain and characteristics, joint sounds, and headache was used.
Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) Axis I Clinical Examination Form questionnaire | A single point in time (1 day)
  Clinical Examination form assesses the site of pain, incisal relationships, mouth opening position, mouth opening and closing movements, lateral and protrusive movements, jaw noise, joint locking, and evaluation of muscle and joint pain by palpation.

SECONDARY OUTCOMES:
The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | A single point in time (1 day)
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) was used to assess the disease activity.
Bath Ankylosing Spondylitis Functional Index (BASFI) | A single point in time (1 day)
  Bath Ankylosing Spondylitis Functional Index (BASFI) is a tool used to assess the functional ability of patients with ankylosing spondylitis. It includes questions about the patient's ability to perform daily activities such as dressing, grooming, standing, and bending.
The Bath Ankylosing Spondylitis Metrology Index (BASMI) | A single point in time (1 day)
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) was used to assess spinal mobility. The Bath Ankylosing Spondylitis Metrology Index (BASMI) includes measurements of tragus-to-wall distance, intermalleolar distance, modified Schober's test, lateral flexion, and cervical rotation.
DC/TMD Axis II-Pain Drawing questionnaire | A single point in time (1 day)
  Pain Drawing which assesses pain location and spread.
DC/TMD Axis II-Patient Health Questionnaire-9 (PHQ-9) | A single point in time (1 day)
  Patient Health Questionnaire-9 (PHQ-9), which assesses depressed mood state.
DC/TMD Axis II- Oral Behaviors Checklist (OBC) | A single point in time (1 day)
  Oral Behaviors Checklist (OBC), which assesses parafunctional behaviors
DC/TMD Axis II-Jaw Functional Limitation Scale-20 (JFLS-20) | A single point in time (1 day)
  Jaw Functional Limitation Scale-20 (JFLS-20) , which assesses limitation of mastication, mobility and verbal end emotional expressions.
DC/TMD Axis II-Patient Health Questionnaire-15 (PHQ-15) | A single point in time (1 day)
  Patient Health Questionnaire-15, which assesses non-specific physical symptoms
DC/TMD Axis II-Graded Chronic Pain Scale; GCPS v2.0 | A single point in time (1 day)
  Graded Chronic Pain Scale (GCPS) is a tool used to assess the severity and impact of chronic pain on a person's life. It involves rating the intensity of pain, as well as how much pain interferes with daily activities and quality of life.
DC/TMD Axis II- General Anxiety Disorder 7 (GAD-7) | A single point in time (1 day)
  The General Anxiety Disorder 7 (GAD-7) is a brief self-report questionnaire that is used to assess the severity of generalized anxiety disorder

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Nur Kesiktaş, Prof, Study Director — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Bilgin E, Bilgin E, Ozdemir O, Kalyoncu U. Temporomandibular disorders in ankylosing spondylitis: a cross-sectional, monocentric study. Rheumatol Int. 2020 Jun;40(6):933-940. doi: 10.1007/s00296-020-04563-y. Epub 2020 Apr 1. PMID 32239320
- [Background] Braun J, Sieper J. Ankylosing spondylitis. Lancet. 2007 Apr 21;369(9570):1379-1390. doi: 10.1016/S0140-6736(07)60635-7. PMID 17448825
- [Background] Huang YF, Chang CT, Muo CH, Chiu KM, Tsai CH, Liu SP. Bidirectional relationship between temporomandibular disorder and ankylosing spondylitis: a population-based cohort study. Clin Oral Investig. 2021 Nov;25(11):6377-6384. doi: 10.1007/s00784-021-03938-0. Epub 2021 Apr 14. PMID 33855657
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Souza RC, de Sousa ET, Sousa D, Sales M, Dos Santos Oliveira R, Mariano MH, Rushansky E, Amorim Gomes AC, Silva E. Prevalence of Temporomandibular Joint Disorders in Patients with Ankylosing Spondylitis: A Cross-Sectional Study. Clin Cosmet Investig Dent. 2021 Nov 11;13:469-478. doi: 10.2147/CCIDE.S320537. eCollection 2021. PMID 34795532
- [Derived] Ahisha BS, Kesiktas FN. Prevalence of temporomandibular joint dysfunction in patients with ankylosing spondylitis and comparison of the findings with healthy controls. Rev Assoc Med Bras (1992). 2024 Sep 30;70(10):e20240807. doi: 10.1590/1806-9282.20240807. eCollection 2024. PMID 39356963